CLINICAL TRIAL: NCT02791438
Title: A Phase 3, Open-label, Multicenter, Long-term Study to Evaluate the Safety, Efficacy and Pharmacokinetics of TAK-536 in Pediatric Patients 6 to Less Than 16 Years of Age With Hypertension
Brief Title: A Phase 3 Long-term Study of TAK-536 in Pediatric Patients 6 to Less Than 16 Years With Hypertension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TAK-536/OCT-101; U1111-1182-4241 (Other: UTN); JapicCTI-163260 (Registry Identifier: JapicCTI)
Record Dates: First submitted 2016-06-01; First posted 2016-06-06 (Estimated); Results first posted 2019-12-23 (Actual); Last update posted 2020-02-07 (Actual); Status verified 2020-02

CONDITIONS: Pediatric Hypertension
MeSH Terms: interventions — azilsartan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Azilsartan 2.5 - 20 mg (Weight < 50 kg) (Experimental): Following a 2-week placebo run-in period, azilsartan 2.5 mg (titrated as needed to the highest dose of 20 mg) was administered orally once daily before or after breakfast, for the participants weighing < 50 kg.
  Interventions: Drug: Azilsartan; Drug: Placebo
- Azilsartan 5 - 40 mg (Weight ≥ 50 kg) (Experimental): Following a 2-week placebo run-in period, azilsartan 5 mg (titrated as needed to the highest dose of 40 mg) was administered orally once daily before or after breakfast, for the participants weighing ≥ 50 kg.
  Interventions: Drug: Azilsartan; Drug: Placebo

INTERVENTIONS:
Drug: Azilsartan — Azilsartan granules and tablets
  Other Names: TAK-536; AZILVA ®
Drug: Placebo — Placebo-matching azilsartan granules and tablets

SUMMARY:
The purpose of this study is to evaluate the safety of administration of azilsartan in pediatric patients aged 6 to less than 16 years with hypertension.

DETAILED DESCRIPTION:
The drug being tested in this study is called azilsartan. Azilsartan is being tested to treat pediatric participants with hypertension.

The study enrolled 27 participants. Following a 2-week Placebo Run-in Period, participants were assigned to one of the two treatment groups based on weight:

* Azilsartan 2.5 - 20 mg (Participants < 50 kg)
* Azilsartan 5 - 40 mg (Participants ≥ 50 kg)

Participants weighing < 50 kg were asked to take an initial dose azilsartan 2.5 mg (titrated as needed to the highest dose of 20 mg) and participants weighing ≥ 50 kg were asked to take an initial dose of 5 mg azilsartan (titrated as needed to the highest dose of 40 mg).

This multi-centre trial was conducted in Japan. The overall time to participate in this study is 56 weeks. The study consisted of a Run-in Period (Week -2 to Week 0), a 52-week Treatment Period, and a 2-week Follow-up Period (up to Week 54). Participants made multiple visits to the clinic and a final visit 2 weeks after the last dose of study drug for follow-up assessment.

ELIGIBILITY:
Inclusion Criteria:

1. In the opinion of the investigator or subinvestigator, the participant's parent or the participant's legal guardian is capable of understanding and complying with protocol requirements.
2. The participant's parent or the participant's legal guardian is capable of signing and dating a written, informed consent form on behalf of the participant prior to the initiation of any study procedures. Written informed assent is also obtained from the participant as much as possible.
3. The Japanese participant who has a diagnosis of hypertension. A participant is eligible if he/she is deemed hypertensive according to the Reference Blood Pressure Values of Children by Gender and Age; office sitting diastolic or systolic blood pressure ≥ 95 percentile for essential hypertension without concomitant hypertensive organ damage, and ≥ 90 percentile for secondary hypertension with concomitant chronic kidney disease (CKD), diabetes mellitus, heart failure or any hypertensive organ damage.

   In addition, participants need to meet the following criteria:

   - If currently treated with any antihypertensive drugs at the start of the Run-in Period: Participant has a documented historical diagnosis of hypertension and an office sitting diastolic or systolic blood pressure meeting the above criteria at the end of the Run-in Period (Week 0).

   - If currently untreated with any antihypertensive drugs at the start of the Run-in Period: Participant who meets the above criteria on 3 separate time points including screening and the end of the Run-in Period (Week 0). In addition, participant with essential hypertension without concomitant hypertensive organ damage still maintains hypertension with non-pharmacotherapy including foods or exercises for at least 3 months within 1 year prior to the start of screening.
4. The participant is male or female and aged 6 to less than 16 years at the time of informed consent.
5. The participant weighs at least 20 kg at screening.
6. The participant is capable of taking the tablets or granules supplied as the study drug.
7. A participant who has undergone kidney transplantation is eligible if he/she underwent the transplantation at least 6 months earlier at screening, and the graft has been functionally stable (estimated glomerular filtration rate (eGFR) ≥ 30 mL/min/1.73 m^2) for at least 6 months with evidence (eg, Doppler echography, computed tomography (CT) scan or magnetic resonance imaging (MRI) excluding grafted kidney arterial stenosis. A participant on immunosuppressive therapy with a stable dose at least 30 days prior to screening is eligible.
8. A female participant of childbearing potential who is sexually active with a nonsterilized male partner agrees to use routinely adequate contraception from signing of informed consent through 1 month after the completion of the study, and proves negative in the pregnancy test at screening.
9. The participants judged by the investigator or subinvestigator that he/she can discontinue the therapy with renin-angiotensin-system (RAS) inhibitors for 2 weeks (acceptable range, 1 to 4 weeks) in safe prior to the Treatment Period.

Exclusion Criteria:

1. The participant has received any investigational compound within 30 days prior to screening or is participating in another clinical study or a post-marketing clinical study.

   Note: This does not apply to participants participating in observational studies without interventional or invasive therapy.
2. The participant previously received therapy with azilsartan. Note: This does not apply to participants participating in single dose pharmacokinetic studies of TAK-536.
3. The participant has poorly controlled hypertension indicated by an office sitting systolic blood pressure higher by at least 15 mmHg and/or an office sitting diastolic blood pressure higher by at least 10 mmHg than the 99 percentiles of the Reference Blood Pressure Values of Children by Gender and Age.
4. The participant has a diagnosis of malignant or accelerated hypertension.
5. The participant was noncompliant (< 70% or > 130%) with the study drug during the Run-in Period.
6. The participant has severe renal dysfunction (eGFR < 30 mL/min/1.73 m^2), is receiving dialysis, has a renovascular disease affecting one or both kidneys, severe nephrotic syndrome not in remission, or a serum albumin level < 2.5 g/dL.
7. The participant has a history of, or the signs/symptoms of serious cardiovascular, hepatobiliary, gastrointestinal, endocrine (eg, hyperthyroidism, Cushing's syndrome), hematological, immunological, urinogenital, psychiatric disease, cancer, or any other disease that adversely affects participant's health, or, in the opinion of the investigator or subinvestigator, potentially confounds the study results.
8. The participant has hemodynamically significant left ventricular outflow obstruction due to aortic stenosis or aortic valvular disease, or is scheduled to undergo a medical procedure affecting blood pressure during the study (eg, correction of arterial anomaly).
9. The participant has a history of or concurrent clinically significant abnormality of 12-lead electrocardiogram (ECG) that, in the opinion of the investigator or subinvestigator, disqualifies the participant for participation in the study.
10. The participant has poorly controlled diabetes mellitus indicated by hemoglobin A1c (HbA1c) > 9.0% at screening.
11. The participant has an alanine aminotransferase (ALT) or aspartate aminotransferase (AST) level ≥ 2.5 × the upper limit of normal (ULN), or a total bilirubin level ≥ 1.5 × ULN at screening, severely impaired hepatic function, any active liver disease (regardless of the cause), or jaundice.
12. The participant has hyperkalemia exceeding ULN at screening.
13. The participant has a history of hepatitis B, hepatitis C, or human immunodeficiency virus (HIV) infection at screening.
14. The participant has a known hypersensitivity or allergy to any angiotensin II receptor blocker (ARBs).
15. The participant needs treatment with any of the excluded medication.
16. If female, the participant is pregnant or lactating or intending to become pregnant before, during, or within 1 month after the completion of this study.

Ages: 6 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 27 (Actual)
Dates: Start 2016-08-18 (Actual); Primary Completion 2019-06-04 (Actual); Study Completion 2019-06-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (30):
- Japan (30):
  - Nagakute, Aichi-ken
  - Nagoya, Aichi-ken
  - Ōbu, Aichi-ken
  - Sapporo, Hokkaido
  - Kobe, Hyōgo
  - Kanazawa, Ishikawa-ken
  - Yokohama, Kanagawa
  - Nankoku, Kochi
  - Sendai, Miyagi
  - Shimajiri-gun, Okinawa
  - Izumi, Osaka
  - Ōsaka-sayama, Osaka
  - Ōtsu, Shiga
  - Shimotsuke, Tochigi
  - Fuchū, Tokyo
  - Nerima-ku, Tokyo
  - Ōta-ku, Tokyo
  - Setagaya-ku, Tokyo
  - Shinjuku-ku, Tokyo
  - Akita
  - Chiba
  - Fukuoka
  - Fukushima
  - Hiroshima
  - Niigata
  - Okayama
  - Osaka
  - Saitama
  - Shizuoka
  - Wakayama

IPD SHARING:
Plan to Share IPD: Yes
Takeda makes patient-level, de-identified data sets and associated documents available for all interventional studies after applicable marketing approvals and commercial availability have been received (or program is completely terminated), an opportunity for the primary publication of the research and final report development has been allowed, and other criteria have been met as set forth in Takeda's Data Sharing Policy (see www.TakedaClinicalTrials.com for details). To obtain access, researchers must submit a legitimate academic research proposal for adjudication by an independent review panel, who will review the scientific merit of the research and the requestor's qualifications and conflict of interest that can result in potential bias. Once approved, qualified researchers who sign a data sharing agreement are provided access to these data in a secure research environment.

REFERENCES:
- See also: Guidelines for Drug Therapy in Pediatric Patients with Cardiovascular Diseases by the Japanese Circulation Society JCS 2012 (JCS 2012) — http://www.j-circ.or.jp/english/cj/index.php/jcs-guidelines/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 17 investigative sites in Japan from 18 August 2016 to 04 June 2019.
Pre-assignment Details: Following a placebo run-in period, pediatric patients with hypertension received azilsartan at starting doses of 2.5 mg for patients < 50 kilograms (kg) and 5 mg for patients ≥ 50 kg.
Period: Run-In Period
Arm/Group | Azilsartan 2.5 - 20 mg (Weight < 50 kg) | Azilsartan 5 - 40 mg (Weight ≥ 50 kg)
Started | 22 | 5
Completed | 22 | 5
Not Completed | 0 | 0
Period: Treatment Period
Arm/Group | Azilsartan 2.5 - 20 mg (Weight < 50 kg) | Azilsartan 5 - 40 mg (Weight ≥ 50 kg)
Started | 22 | 5
Completed | 19 | 4
Not Completed | 3 | 1
Not completed — Adverse Event | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Withdrawal by Parent/Guardian | 2 | 0

BASELINE CHARACTERISTICS:
Population: Safety analysis set included all randomized participants who received at least 1 dose of the study drug for the Treatment Period.
Groups:
- Total: Total of all reporting groups
Arm/Group | Azilsartan 2.5 - 20 mg (Weight < 50 kg) | Azilsartan 5 - 40 mg (Weight ≥ 50 kg) | Total
Number analyzed (Participants) | 22 | 5 | 27
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.0 (2.54) | 12.8 (2.49) | 9.7 (2.91)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 1 | 10
  Male | 13 | 4 | 17
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Japan | 22 | 5 | 27
Height [Mean (Standard Deviation); unit: cm] | 128.4 (10.92) | 160.4 (16.30) | 134.3 (17.26)
Weight [Mean (Standard Deviation); unit: kg] | 31.94 (8.306) | 63.78 (10.139) | 37.83 (15.180)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — BMI is participants weight in kilograms (kg) divided by his or her height in meters squared (m^2).
  kg/m^2 | 19.29 (4.216) | 24.86 (2.726) | 20.32 (4.513)
Disease Duration [Mean (Standard Deviation); unit: years] | 2.30 (2.152) | 1.66 (2.418) | 2.18 (2.168)
Office Sitting Blood Pressure (Systolic) at Week 0 [Mean (Standard Deviation); unit: mmHg] — Office trough sitting blood pressure is defined as the blood pressure collected in the office while the participant was sitting at a time point immediately before dosing.
  mmHg | 123.2 (12.55) | 136.6 (8.32) | 125.7 (12.89)
Office Sitting Blood Pressure (Diastolic) at Week 0 [Mean (Standard Deviation); unit: mmHg] — Office trough sitting blood pressure is defined as the blood pressure collected in the office while the participant was sitting at a time point immediately before dosing.
  mmHg | 72.1 (14.01) | 71.6 (11.87) | 72.0 (13.43)
Estimated Glomerular Filtration Rate (eGFR) [Mean (Standard Deviation); unit: mL/min/1.73m^2] | 99.571 (30.9858) | 131.438 (26.1758) | 105.472 (32.2493)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Reporting One or More Treatment-emergent Adverse Events (TEAEs)
Description: An Adverse Event (AE) is defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (eg, a clinically significant abnormal laboratory finding), symptom, or disease temporally associated with the use of a drug, whether or not it is considered related to the drug. A treatment-emergent adverse event (TEAE) is defined as an adverse event with an onset that occurs or worsens after receiving study drug.
Time Frame: Up to Week 54
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Azilsartan 2.5 - 20 mg (Weight < 50 kg) | Azilsartan 5 - 40 mg (Weight ≥ 50 kg)
Number analyzed (Participants) | 22 | 5
Participants | 19 | 5

2. Primary Outcome: Number of Participants With TEAEs Related to Anthropometric Measurement (Weight, Height and Body Mass Index (BMI))
Description: as for outcome 1
Time Frame: Up to Week 54
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Azilsartan 2.5 - 20 mg (Weight < 50 kg) | Azilsartan 5 - 40 mg (Weight ≥ 50 kg)
Number analyzed (Participants) | 22 | 5
Participants | 0 | 0

3. Primary Outcome: Number Of Participants With Markedly Abnormal Values of Laboratory Parameters
Description: The laboratory values outside the range (Blood Urea Nitrogen (BUN) (mg/dL) >30, Creatinine (mg/dL) >2.0, eGFR (mL/min/1.73m^2) <30, Creatine Kinase (U/L) >5×ULN) are considered markedly abnormal.
Time Frame: Up to Week 54
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Azilsartan 2.5 - 20 mg (Weight < 50 kg) | Azilsartan 5 - 40 mg (Weight ≥ 50 kg)
Number analyzed (Participants) | 22 | 5
Participants
  Blood Urea Nitrogen (BUN) (mg/dL) >30 | 2 | 1
  Creatinine (mg/dL) >2.0 | 1 | 0
  eGFR (mL/min/1.73m^2) <30 | 1 | 0
  Creatine Kinase (U/L) >5×ULN | 0 | 1

4. Primary Outcome: Number Of Participants With TEAEs Related To Resting 12-Lead Electrocardiogram (ECG)
Description: A standard 12-lead ECG was performed while the participant was at rest. Any abnormal ECG findings determined by the investigator to be clinically significant were reported as adverse events.
Time Frame: Up to Week 54
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Azilsartan 2.5 - 20 mg (Weight < 50 kg) | Azilsartan 5 - 40 mg (Weight ≥ 50 kg)
Number analyzed (Participants) | 22 | 5
Participants | 0 | 0

5. Primary Outcome: Number Of Participants With TEAEs Related To Vital Signs (Hypotension)
Description: A treatment-emergent adverse event (TEAE) is defined as an adverse event with an onset that occurs after receiving study drug. Vital signs included office standing blood pressure, office sitting pulse rate, office standing pulse rate, and home sitting blood pressure. Any abnormal vital signs findings determined by the investigator to be clinically significant were reported as adverse events.
Time Frame: Up to Week 54
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Azilsartan 2.5 - 20 mg (Weight < 50 kg) | Azilsartan 5 - 40 mg (Weight ≥ 50 kg)
Number analyzed (Participants) | 22 | 5
Participants | 1 | 0

6. Secondary Outcome: Change From Baseline in Office Trough Sitting Systolic Blood Pressure
Description: Office trough sitting blood pressure is defined as the blood pressure collected in the office while the participant was sitting at a time point immediately before the next dosing, when the blood drug concentration is assumed to be the lowest. A negative change from Baseline indicates improvement. The data of change from baseline to the End of Treatment Period I (EOT 1) and the End of the Treatment Period 2 (EOT 2) were calculated with the evaluable data within the acceptable time points (EOT1 was for up to Week 12 and EOT2 was for up to Week 52) with the largest Study Day was used. Meanwhile, change from baseline to Week 12 and 52 were calculated with the data of Week 12 and 52 respectively.
Time Frame: Baseline (Day 0), Weeks 2, 4, 8, 12,16, 20, 24, 32, 40, 52, Week 54 (Follow-up), End-of-treatment (EOT) 1 (Up to Week 12), EOT 2 (Up to Week 52)
Population: Full analysis set included all the randomized participants. Number analyzed is the number of participants with data available at the given timepoint for this outcome measure.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Azilsartan 2.5 - 20 mg (Weight < 50 kg) | Azilsartan 5 - 40 mg (Weight ≥ 50 kg)
Number analyzed (Participants) | 22 | 5
mmHg
  Change from Baseline at Week 2 | -7.8 (11.34) | -7.4 (5.68)
  Change from Baseline at Week 4 | -10.7 (12.64) | -13.2 (11.43)
  Change from Baseline at Week 8 | -10.1 (10.41) | -13.0 (10.12)
  Change from Baseline at Week 12: number analyzed (Participants) | 19 | 5
  Change from Baseline at Week 12 | -13.0 (10.30) | -7.6 (10.21)
  Change from Baseline at Week 16: number analyzed (Participants) | 21 | 5
  Change from Baseline at Week 16 | -13.1 (12.61) | -17.6 (6.58)
  Change from Baseline at Week 20: number analyzed (Participants) | 21 | 5
  Change from Baseline at Week 20 | -10.0 (11.23) | -16.6 (11.22)
  Change from Baseline at Week 24: number analyzed (Participants) | 20 | 5
  Change from Baseline at Week 24 | -12.9 (13.95) | -9.4 (11.97)
  Change from Baseline at Week 32: number analyzed (Participants) | 20 | 4
  Change from Baseline at Week 32 | -13.6 (16.29) | -15.3 (10.90)
  Change from Baseline at Week 40: number analyzed (Participants) | 20 | 4
  Change from Baseline at Week 40 | -10.3 (14.32) | -17.5 (12.61)
  Change from Baseline (BL) at Week 52: number analyzed (Participants) | 19 | 4
  Change from Baseline (BL) at Week 52 | -8.9 (12.29) | -17.5 (8.89)
  Change from BL at Week 54 Follow-up: number analyzed (Participants) | 17 | 2
  Change from BL at Week 54 Follow-up | -4.4 (12.65) | -14.5 (2.12)
  Change from BL at EOT 1 (Up to Week 12) | -13.5 (10.27) | -7.6 (10.21)
  Change from BL at EOT 2 (Up to Week 52) | -8.8 (11.79) | -15.4 (9.02)

7. Secondary Outcome: Change From Baseline in Office Trough Sitting Diastolic Blood Pressure
Description: as for outcome 6
Time Frame: Baseline (Day 0), Weeks 2, 4, 8, 12,16, 20, 24, 32, 40, 52, Week 54 (Follow-up), EOT 1 (Up to Week 12), EOT 2 (Up to Week 52)
Population: Full analysis set included all the randomized participants. Number analyzed is the number participants with data available at the given timepoint for this outcome measure.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Azilsartan 2.5 - 20 mg (Weight < 50 kg) | Azilsartan 5 - 40 mg (Weight ≥ 50 kg)
Number analyzed (Participants) | 22 | 5
mmHg
  Change from Baseline at Week 2 | -7.5 (11.81) | -9.8 (5.63)
  Change from Baseline at Week 4 | -11.5 (14.11) | -11.2 (10.21)
  Change from Baseline at Week 8 | -11.8 (13.06) | -11.6 (11.01)
  Change from Baseline at Week 12: number analyzed (Participants) | 19 | 5
  Change from Baseline at Week 12 | -14.0 (13.30) | -10.0 (10.77)
  Change from Baseline at Week 16: number analyzed (Participants) | 21 | 5
  Change from Baseline at Week 16 | -13.4 (13.79) | -16.6 (8.08)
  Change from Baseline at Week 20: number analyzed (Participants) | 21 | 5
  Change from Baseline at Week 20 | -13.5 (13.87) | -13.8 (9.78)
  Change from Baseline at Week 24: number analyzed (Participants) | 20 | 5
  Change from Baseline at Week 24 | -14.1 (16.04) | -10.8 (7.79)
  Change from Baseline at Week 32: number analyzed (Participants) | 20 | 4
  Change from Baseline at Week 32 | -11.4 (15.51) | -15.8 (15.90)
  Change from Baseline at Week 40: number analyzed (Participants) | 20 | 4
  Change from Baseline at Week 40 | -11.2 (16.47) | -12.0 (11.69)
  Change from Baseline (BL) at Week 52: number analyzed (Participants) | 19 | 4
  Change from Baseline (BL) at Week 52 | -10.7 (14.50) | -15.3 (10.81)
  Change from BL at Week 54 Follow-up: number analyzed (Participants) | 17 | 2
  Change from BL at Week 54 Follow-up | -6.1 (9.97) | -14.0 (5.66)
  Change from BL at EOT I (Up to Week 12) | -14.8 (13.80) | -10.0 (10.77)
  Change from BL at EOT 2 (Up to Week 52) | -10.3 (13.97) | -13.6 (10.06)

8. Secondary Outcome: Percentage Of Participants Who Achieve The Target Blood Pressure
Description: Target blood pressure is defined as the normal reference range for blood pressure by age according to Guidelines for Drug Therapy in Pediatric Patients with Cardiovascular Diseases by the Japanese Circulation Society JCS 2012 (JCS 2012). The data of change from baseline to EOT 1 and EOT 2 were calculated with the evaluable data within the acceptable time points (EOT1 was for up to Week 12 and EOT2 was for up to Week 52) with the largest Study Day was used. Meanwhile, change from baseline to Week 12 and 52 were calculated with the data of Week 12 and 52 respectively. Target blood pressure were described on Guidelines for Drug Therapy in Pediatric Patients with Cardiovascular Diseases by the Japanese Circulation Society JCS 2012 (JCS 2012) (see Links on Registration Section).
Time Frame: Weeks 2, 4, 8, 12,16, 20, 24, 32, 40, 52, Week 54 (Follow-up), EOT 1 (Up to Week 12), EOT 2 (Up to Week 52)
Population: as for outcome 6
Measure: Number; unit: percentage of participants
Arm/Group | Azilsartan 2.5 - 20 mg (Weight < 50 kg) | Azilsartan 5 - 40 mg (Weight ≥ 50 kg)
Number analyzed (Participants) | 22 | 5
percentage of participants
  Week 2 | 45.5 | 40.0
  Week 4 | 45.5 | 20.0
  Week 8 | 50.0 | 60.0
  Week 12: number analyzed (Participants) | 19 | 5
  Week 12 | 73.7 | 40.0
  Week 16: number analyzed (Participants) | 21 | 5
  Week 16 | 66.7 | 40.0
  Week 20: number analyzed (Participants) | 21 | 5
  Week 20 | 57.1 | 40.0
  Week 24: number analyzed (Participants) | 20 | 5
  Week 24 | 50.0 | 20.0
  Week 32: number analyzed (Participants) | 20 | 4
  Week 32 | 50.0 | 75.0
  Week 40: number analyzed (Participants) | 20 | 4
  Week 40 | 45.0 | 75.0
  Week 52: number analyzed (Participants) | 19 | 4
  Week 52 | 36.8 | 75.0
  Week 54 (Follow-up): number analyzed (Participants) | 17 | 2
  Week 54 (Follow-up) | 41.2 | 50.0
  EOT 1 (Up to Week 12) | 68.2 | 40.0
  EOT 2 (Up to Week 52) | 36.4 | 60.0

9. Secondary Outcome: Observed Plasma Concentration for Azilsartan
Description: Reported data were observed plasma concentration for Azilsartan for each arm. Dosage of the study drug after Week 2 (postdose) is different among participants.
Time Frame: Predose and 2 hours postdose Weeks 2, 4, 8, 12 and 2 hours postdose Week 16
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: ug/L
Arm/Group | Azilsartan 2.5 - 20 mg (Weight < 50 kg) | Azilsartan 5 - 40 mg (Weight ≥ 50 kg)
Number analyzed (Participants) | 22 | 5
ug/L
  Week 2 (Predose): number analyzed (Participants) | 20 | 5
  Week 2 (Predose) | 22.3 (18.64) | 16.8 (10.50)
  Week 2 (Postdose): number analyzed (Participants) | 4 | 2
  Week 2 (Postdose) | 206.0 (157.18) | 610.0 (12.73)
  Week 4 (Predose): number analyzed (Participants) | 21 | 4
  Week 4 (Predose) | 31.1 (23.35) | 35.0 (19.66)
  Week 4 (Postdose): number analyzed (Participants) | 2 | 1
  Week 4 (Postdose) | 175.0 (125.87) | 64.0 (NA) — Standard deviation was not calculated for 1 participant.
  Week 8 (Predose): number analyzed (Participants) | 18 | 1
  Week 8 (Predose) | 49.2 (60.74) | 58.0 (31.65)
  Week 8 (Postdose): number analyzed (Participants) | 2 | 1
  Week 8 (Postdose) | 221.5 (177.48) | 587.0 (NA) — Standard deviation was not calculated for 1 participant.
  Week 12 (Predose): number analyzed (Participants) | 19 | 4
  Week 12 (Predose) | 48.9 (55.01) | 64.8 (37.83)
  Week 12 (Postdose): number analyzed (Participants) | 1 | 1
  Week 12 (Postdose) | 802.0 (NA) — Standard deviation was not calculated for 1 participant. | 116.0 (NA) — Standard deviation was not calculated for 1 participant.
  Week 16 (Postdose): number analyzed (Participants) | 21 | 5
  Week 16 (Postdose) | 743.1 (590.29) | 1675.8 (1579.32)

10. Secondary Outcome: Observed Plasma Concentration for Azilsartan Metabolites (M-I)
Description: Reported data were observed plasma concentration for Azilsartan Metabolites (M-I) for each arm. Dosage of the study drug after Week 2 (postdose) is different among participants.
Time Frame: Predose and 2 hours postdose Weeks 2, 4, 8, 12 and 2 hours postdose Week 16
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: ug/L
Arm/Group | Azilsartan 2.5 - 20 mg (Weight < 50 kg) | Azilsartan 5 - 40 mg (Weight ≥ 50 kg)
Number analyzed (Participants) | 22 | 5
ug/L
  Week 2 (Predose): number analyzed (Participants) | 20 | 5
  Week 2 (Predose) | 1.9 (2.15) | 1.4 (1.14)
  Week 2 (Postdose): number analyzed (Participants) | 4 | 2
  Week 2 (Postdose) | 16.3 (9.54) | 21.0 (1.41)
  Week 4 (Predose): number analyzed (Participants) | 21 | 4
  Week 4 (Predose) | 2.7 (2.92) | 3.3 (2.63)
  Week 4 (Postdose): number analyzed (Participants) | 2 | 1
  Week 4 (Postdose) | 6.5 (6.36) | 4.0 (NA) — Standard deviation was not calculated for 1 participant.
  Week 8 (Predose): number analyzed (Participants) | 18 | 4
  Week 8 (Predose) | 3.1 (3.33) | 3.8 (2.36)
  Week 8 (Postdose): number analyzed (Participants) | 2 | 1
  Week 8 (Postdose) | 37.5 (21.92) | 25.0 (NA) — Standard deviation was not calculated for 1 participant.
  Week 12 (Predose): number analyzed (Participants) | 19 | 4
  Week 12 (Predose) | 3.6 (3.36) | 7.5 (5.69)
  Week 12 (Postdose): number analyzed (Participants) | 1 | 1
  Week 12 (Postdose) | 51.0 (NA) — Standard deviation was not calculated for 1 participant. | 4.0 (NA) — Standard deviation was not calculated for 1 participant.
  Week 16 (Postdose): number analyzed (Participants) | 21 | 5
  Week 16 (Postdose) | 39.2 (30.60) | 59.8 (40.07)

11. Secondary Outcome: Observed Plasma Concentration for Azilsartan Metabolites (M-II)
Description: Reported data were observed plasma concentration for Azilsartan Metabolites (M-II) for each arm. Dosage of the study drug after Week 2 (postdose) is different among participants.
Time Frame: Predose and 2 hours postdose Weeks 2, 4, 8, 12 and 2 hours postdose Week 16
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: ug/L
Arm/Group | Azilsartan 2.5 - 20 mg (Weight < 50 kg) | Azilsartan 5 - 40 mg (Weight ≥ 50 kg)
Number analyzed (Participants) | 22 | 5
ug/L
  Week 2 (Predose): number analyzed (Participants) | 20 | 5
  Week 2 (Predose) | 53.3 (61.31) | 41.4 (28.66)
  Week 2 (Postdose): number analyzed (Participants) | 4 | 2
  Week 2 (Postdose) | 158.3 (102.88) | 129.0 (26.87)
  Week 4 (Predose): number analyzed (Participants) | 21 | 4
  Week 4 (Predose) | 71.1 (77.05) | 90.8 (40.99)
  Week 4 (Postdose): number analyzed (Participants) | 2 | 1
  Week 4 (Postdose) | 186.0 (214.96) | 69 (NA) — Standard deviation was not calculated for 1 participant.
  Week 8 (Predose): number analyzed (Participants) | 18 | 4
  Week 8 (Predose) | 113.8 (140.23) | 124.0 (78.25)
  Week 8 (Postdose): number analyzed (Participants) | 2 | 1
  Week 8 (Postdose) | 175.5 (78.49) | 110.0 (NA) — Standard deviation was not calculated for 1 participant.
  Week 12 (Predose): number analyzed (Participants) | 19 | 4
  Week 12 (Predose) | 106.2 (144.85) | 180.0 (147.97)
  Week 12 (Postdose): number analyzed (Participants) | 1 | 1
  Week 12 (Postdose) | 184.0 (NA) — Standard deviation was not calculated for 1 participant. | 86.0 (NA) — Standard deviation was not calculated for 1 participant.
  Week 16 (Postdose): number analyzed (Participants) | 21 | 5
  Week 16 (Postdose) | 311.0 (480.62) | 423.6 (277.62)

ADVERSE EVENTS:
Time Frame: From the first dose of study drug up to last dose of study drug plus 2 weeks (up to 62 Weeks)
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment. The safety population (SAF) includes all randomized participants who received at least 1 dose of study medication in treatment period.
Arm/Group | Azilsartan 2.5 - 20 mg (Weight < 50 kg) | Azilsartan 5 - 40 mg (Weight ≥ 50 kg)
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/5
Serious Adverse Events (participants affected / at risk) | 2/22 | 0/5
Other Adverse Events (participants affected / at risk) | 19/22 | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Azilsartan 2.5 - 20 mg (Weight < 50 kg) (N=22) | Azilsartan 5 - 40 mg (Weight ≥ 50 kg) (N=5)
Kidney transplant rejection (Immune system disorders) | 1 | 0
Varicella (Infections and infestations) | 1 | 0
Complications of transplanted kidney (Injury, poisoning and procedural complications) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Azilsartan 2.5 - 20 mg (Weight < 50 kg) (N=22) | Azilsartan 5 - 40 mg (Weight ≥ 50 kg) (N=5)
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 1 | 0
Nephrogenic anaemia (Blood and lymphatic system disorders) | 1 | 0
Dry eye (Eye disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 3 | 1
Abdominal pain (Gastrointestinal disorders) | 3 | 0
Stomatitis (Gastrointestinal disorders) | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Enteritis (Gastrointestinal disorders) | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Pyrexia (General disorders) | 3 | 0
Chest pain (General disorders) | 1 | 0
Malaise (General disorders) | 1 | 0
Vessel puncture site bruise (General disorders) | 1 | 0
Seasonal allergy (Immune system disorders) | 1 | 0
Nasopharyngitis (Infections and infestations) | 9 | 2
Gastroenteritis (Infections and infestations) | 4 | 0
Influenza (Infections and infestations) | 3 | 1
Otitis media (Infections and infestations) | 3 | 0
Sinusitis (Infections and infestations) | 2 | 0
Upper respiratory tract infection (Infections and infestations) | 2 | 0
Adenoiditis (Infections and infestations) | 1 | 0
Adenovirus infection (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 1 | 0
Conjunctivitis (Infections and infestations) | 1 | 0
Coxsackie viral infection (Infections and infestations) | 1 | 0
Lice infestation (Infections and infestations) | 1 | 0
Hordeolum (Infections and infestations) | 1 | 0
Mumps (Infections and infestations) | 1 | 0
Parotitis (Infections and infestations) | 1 | 0
Pharyngitis (Infections and infestations) | 0 | 1
Rhinitis (Infections and infestations) | 0 | 1
Streptococcal infection (Infections and infestations) | 1 | 0
Tinea manuum (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 2 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 2 | 0
Ear injury (Injury, poisoning and procedural complications) | 1 | 0
Heat stroke (Injury, poisoning and procedural complications) | 1 | 0
Human bite (Injury, poisoning and procedural complications) | 1 | 0
Ligament injury (Injury, poisoning and procedural complications) | 1 | 0
Blood creatinine increased (Investigations) | 2 | 0
Protein urine present (Investigations) | 1 | 0
White blood cell count increased (Investigations) | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Dizziness (Nervous system disorders) | 3 | 0
Headache (Nervous system disorders) | 3 | 0
Dizziness postural (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 0 | 1
Renal impairment (Renal and urinary disorders) | 1 | 1
Dysuria (Renal and urinary disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal obstruction (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Acne (Skin and subcutaneous tissue disorders) | 1 | 0
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 2 | 0
Eczema (Skin and subcutaneous tissue disorders) | 1 | 0
Eczema asteatotic (Skin and subcutaneous tissue disorders) | 1 | 0
Leukoderma (Skin and subcutaneous tissue disorders) | 1 | 0
Skin erosion (Skin and subcutaneous tissue disorders) | 0 | 1
Solar dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0
Hypotension (Vascular disorders) | 1 | 0
Orthostatic hypotension (Vascular disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.

DOCUMENTS (2):
  • Study Protocol (2017-04-12): https://cdn.clinicaltrials.gov/large-docs/38/NCT02791438/Prot_000.pdf
  • Statistical Analysis Plan (2018-10-05): https://cdn.clinicaltrials.gov/large-docs/38/NCT02791438/SAP_001.pdf